CLINICAL TRIAL: NCT01366222
Title: Food Concentrates Supplementation to Alleviate Asthma in Children
Acronym: FSAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academia Sinica, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Wen-Harn Pan, Principal investigator, Academia Sinica, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AS-IRB02- 07022
Record Dates: First submitted 2011-05-25; First posted 2011-06-06 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma | interventions — Vegetables; Fish Oils; Probiotics; Fruit

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: food concentrates: fruit, vegetable, fish oil and probiotics
- Food concentrates (FC) (Active Comparator): Food concentrates (FC) was including fruit and vegetable, fish and probiotics.
  Interventions: Dietary Supplement: food concentrates: fruit, vegetable, fish oil and probiotics

INTERVENTIONS:
Dietary Supplement: food concentrates: fruit, vegetable, fish oil and probiotics — comparison the effect of food concentrate
  Other Names: fruit and vegetable concentrates; fish oil; probiotics

SUMMARY:
The purpose of this study is to determine whether food concentrates supplementation (vegetable plus fruit, fish, probiotics) are effective to alleviate drug used, asthma symptoms and lung function in children due to asthma.

DETAILED DESCRIPTION:
The prevalence of asthma is increasing in Taiwan and worldwide. This could be related to dietary factors and their interactions with genes and the environment. Ample evidence from cross-sectional and case-control observational studies suggested that consumption level of fruits, vegetables, and potentially vitamins A, C, E from foods have negative association with asthma risk, and positive association with lung function. However, single nutrient supplementation neither improved asthma symptoms and lung function, nor reduced inflammatory mediators. Some studies had shown probiotics could regulate human immunity. A number of trials have suggested that fish oil supplement improves lung function and reduces inflammatory mediator. The potential interactions among multiple components in foods have been neglected in the past. Recently, observational studies on dietary pattern analyses or intervention trials modifying the overall dietary composition have caught tremendous scientific attentions. Therefore, the investigators will design an intervention trial with food-based principle to investigate the the joint effect of several beneficial dietary components on asthma symptoms. For practicality and efficiency, vegetable plus fruit concentrates, fish oil, and probiotic concentrate are considered as supplements to asthmatic children. The investigators hope that the study can provided a direction for dietary modification in asthma children.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma

Exclusion Criteria:

* subjects received immunotherapy over the past 6 months
* Long-term used oral corticosteroids
* have other diseases such as heart disease, kidney disease, liver abnormalities
* have been supplement fish oil, probiotics, and high levels of vitamin supplements in the past three months
* vegetarian
* subjects have hemorrhagic disease

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The change of pediatric asthma quality of life questionnaire score (PAQLQ score) at three time points | Baseline, 8 weeks and 16 weeks after intervention

SECONDARY OUTCOMES:
The change of pulmonary functions (FVC, FEV1) at three time points | Baseline, 8weeks and 16 weeks after intervention
The change of medicine usage at three time points | Baseline, 8 weeks and 16 weeks after intervention
The change of asthma control test score(ACT) at three time points | Baseline, 4, 8,12 and 16 weeks after intervention
weekly diary | Baseline and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15 and 16 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Han Pan, Ph. D., Principal Investigator — Academia Sinica, Taiwan
Locations (1):
- Academia Sinica, Taipei, Taiwan